CLINICAL TRIAL: NCT00821080
Title: A Phase I Study of Vandetanib and Sirolimus in Patients With Recurrent Glioblastoma
Brief Title: Vandetanib and Sirolimus in Patients With Recurrent Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Dana-Farber Cancer Institute (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Tracy T. Batchelor, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-396
Record Dates: First submitted 2009-01-09; First posted 2009-01-13 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Glioblastoma
Keywords: vandetanib; sirolimus; recurrent glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Sirolimus; vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vandetanib and Sirolimus (Experimental): Single arm study
  Interventions: Drug: Sirolimus; Drug: Vandetanib

INTERVENTIONS:
Drug: Sirolimus — Taken orally at different dose levels depending upon enrollment time period
Drug: Vandetanib — Taken orally at different dose levels depending upon enrollment time period

SUMMARY:
This study is evaluating a combination of drugs called sirolimus and vandetanib to treat glioblastoma. Sirolimus has been approved for use in patients who undergo organ transplants. Sirolimus works by suppressing the immune system so the body will not reject the transplanted organ. Vandetanib is an investigational drug and we are trying to find the highest and safest dose of vandetanib with sirolimus that can be given safely.

DETAILED DESCRIPTION:
* Vandetanib will be given to participants in tablet form. The dose taken will depend upon when they are enrolled in the study. The doctor will inform them of which dose they are on and how many tablets they will be taking.
* Sirolimus will also be given to participants in tablet form. The dose taken will depend upon when they are enrolled in the study. The dose on the first day will be higher than the dose taken every other day.
* Participants will also be given Bactrim, one double-strength table three times each week (Monday, Wednesday, Friday) to help prevent participants from getting a type of pneumonia called pneumocystis pneumonia.
* The following tests and procedures will be performed before the participants begin taking the study drugs and before every 4 week cycle: Physical exam; medical history; questions about any side effects; tumor assessment by MRI or CT (only before every other cycle); Mini-Mental Status exam (MMSE); ECG (week 1, 2, 4, 8, 12, then every 3 months thereafter); blood pressure; blood tests and urine tests.
* Participants will be in this research study for a maximum of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma at some point in their disease course
* All patients must have received prior standard therapy including resection if feasible, radiation and temozolomide
* May have received 3 or fewer chemotherapy or biotherapy systemic regimens. Gliadel wafer therapy is not counted as a regimen. Patients may not have received any prior anti-VEGF, anti-EGF therapy or mTOR inhibitors.
* Lab values as outlined in protocol
* Must have recovered from immediate post-operative period and must be maintained on stable or decreasing corticosteroid regimen for at least 3 days prior to the start of treatment
* Must have recovered from possible complications of prior chemotherapies and have a period of 28-42 days since last treatment. Patients must be at least 4 weeks from a non-nitrosourea chemotherapy or 6 weeks from a nitrosourea chemotherapy. Patients must be at least 1 week from the use of non-cytotoxic therapies
* Must be at least 3 months from the completion of radiation or radiosurgery
* Must have documented progression of the disease on the MRI scan using Macdonald criteria
* KPS 60 or greater
* Mini-Mental Status Examination (MMSE) Score > 15
* 18 years of age or older
* All female participants of childbearing potential must have a negative pregnancy test prior to enrollment

Exclusion Criteria:

* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the Investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardize compliance with the protocol
* Clinically significant cardiovascular event within 3 months before entry; or presence of cardiac disease that, in the opinion of the Investigator, increases the risk of ventricular arrhythmia
* History of arrhythmia which is symptomatic or requires treatment or asymptomatic sustained ventricular tachycardia. Atrial fibrillation, controlled on medication is NOT an exclusion
* Previous history of QTc prolongation as a result from other medication that required discontinuation of that medication
* Congenital QTc syndrome or 1st degree relative with unexplained sudden death under 40 years of age
* Presence of left bundle branch block (LBBB)
* QTc with Bazett's correction that is unmeasurable or 480 or greater msec on screening ECG
* Any concomitant medication that may cause QTc prolongation, induce Torsades de Pointes or induce CYP3A4 function
* Hypertension not controlled by medical therapy
* Currently active diarrhea that may affect the ability of the patient to absorb the vandetanib. Specifically, patients with diarrhea of CTCAE v3.0 grade III or above will be excluded
* Women who are currently pregnant or breast-feeding
* Previous or current malignancies of other histologies within the last 5 years, with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
* Receipt of any investigational agents within 30 days prior to commencing study treatment
* Any unresolved toxicity greater than CTC grade 1 from previous anti-cancer therapy
* Major surgery, including craniotomy for tumor resection, within 4 weeks or incompletely healed surgical incision before starting study therapy. Stereotactic biopsy of the tumor within 2 weeks of starting therapy
* Patients on enzyme-inducing anti-epileptic (EIAED) drug therapy
* Patients unable to undergo MRI evaluation prior to potential enrollment
* Patients who, in the opinion of the treating neuro-oncologist, have a significant intratumoral or peritumoral hemorrhage evident on pre-therapy MRI
* Patients with a history of wound-healing disorders, advanced coronary disease, or with a recent history (<1 year) of peptic ulcer disease
* Patients with serious and chronic liver function abnormalities and uncontrolled hyperlipidemia
* Patients unable to be treated with medications for PCP prophylaxis
* Patients with documented allergy to sirolimus
* Patients who are severely immunosuppressed
* Current anticoagulation is NOT criteria for exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-10; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To determine the optimal, safe dose of vandetanib in combination with sirolimus. MTD and dose-limiting toxicity (DLT) of this combination therapy will also be established | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Batchelor, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Instiute, Boston, Massachusetts

REFERENCES:
- [Derived] Chheda MG, Wen PY, Hochberg FH, Chi AS, Drappatz J, Eichler AF, Yang D, Beroukhim R, Norden AD, Gerstner ER, Betensky RA, Batchelor TT. Vandetanib plus sirolimus in adults with recurrent glioblastoma: results of a phase I and dose expansion cohort study. J Neurooncol. 2015 Feb;121(3):627-34. doi: 10.1007/s11060-014-1680-2. Epub 2014 Dec 13. PMID 25503302